CLINICAL TRIAL: NCT06540469
Title: Effects of Optimal Iodine Supplementation in Anti-thyroid Drug Therapy for Graves' Hyperthyroidism: a Prospective Randomized Controlled Trial
Brief Title: Iodine Supplementation in Graves' Hyperthyroidism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: First Hospital of China Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Hai-qing Zhang, Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240521
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Graves Disease; Hyperthyroidism
Keywords: Graves' Disease; Hyperthyroidism; Iodine Supplementation; Anti-Thyroid Drug
MeSH Terms: conditions — Graves Disease; Hyperthyroidism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iodine Supplementation in Whole Course of Treatment with ATDs (Experimental)
  Interventions: Dietary Supplement: Iodine Supplementation in Whole Course of Treatment with ATDs; Drug: anti-Thyroid Drugs
- Iodine Supplementation During Maintenance Treatment with ATDs (Experimental)
  Interventions: Dietary Supplement: Iodine Supplementation During Maintenance Treatment with ATDs; Drug: anti-Thyroid Drugs
- Iodine Restriction in Whole Course of Treatment with ATDs (Other)
  Interventions: Dietary Supplement: Iodine Restriction in Whole Course of Treatment with ATDs; Drug: anti-Thyroid Drugs

INTERVENTIONS:
Dietary Supplement: Iodine Supplementation in Whole Course of Treatment with ATDs — Moderate iodine supplementation (150μg iodine per day, equivalently 7-9g iodized salt per day) will be taken from ATDs treatment starting until 1 year after ATDs withdrawal.
  Arms: Iodine Supplementation in Whole Course of Treatment with ATDs
Dietary Supplement: Iodine Supplementation During Maintenance Treatment with ATDs — Iodine restriction (non-iodized salt and low iodine diet) will be demanded at the early course of ATDs treatment, and moderate iodine supplementation (150μg iodine per day, equivalently 7-9g iodized salt per day) will be taken when the ATDs dose is titrated down to a maintenance level until 1 year after ATDs withdrawal.
  Arms: Iodine Supplementation During Maintenance Treatment with ATDs
Dietary Supplement: Iodine Restriction in Whole Course of Treatment with ATDs — Iodine restriction (non-iodized salt and low iodine diet) will be demanded from ATDs treatment starting until 1 year after ATDs withdrawal.
  Arms: Iodine Restriction in Whole Course of Treatment with ATDs
Drug: anti-Thyroid Drugs — Individualized methimazole (MMI)

SUMMARY:
In China, the morbidity of thyroid diseases is high and the harm is serious. Iodine is closely related to thyroid diseases. It should be paid attention to guide patients to supplement iodine scientifically. Thyroid iodine uptake in hyperthyroidism patients is enhanced, and patients are generally advised to limit iodine intake in clinical practice. However, recent studies suggest that there is no definite conclusion on whether patients with hyperthyroidism should strictly limit iodine intake. The purpose of this study is to establish a national multi-center iodine intervention cohort for patients with Graves' hyperthyroidism, identify the effects of different iodine intake on hyperthyroidism, and establish iodine intervention program for hyperthyroidism. This study is a multicenter, prospective, open-level, randomized, controlled, parallel group clinical trial with a total sample size of 315 cases, a total of 3 participating units, each of which completed 105 cases. All subjects meeting the inclusion criteria were completely randomized in each center according to the random procedure with a probability of 1:1:1: ① Iodine Supplementation in Whole Course of Treatment with ATDs; ② Iodine Supplementation During Maintenance Treatment with ATDs; ③ Iodine Restriction in Whole Course of Treatment with ATDs. Information was collected before ATD treatment, at 3 months, 6 months, 12 months, 18 months (withdrawal), 6 months and 12 months after ATDs withdrawal. The primary purpose of this study is to analyze the difference in remission rate of hyperthyroidism between different iodine nutritional interventions. At the same time, the differences of duration from initiation to withdrawal of ATDs, duration from initiation of ATDs to thyroid function (including serum FT3, FT4 and TSH) normalization, duration from initiation of ATDs to serum FT3 and FT4 normalization, quality of life (QOL) in patients with Graves' hyperthyroidism, adverse effects rate of ATDs treatment, duration from initiation of ATDs to serum negative TRAb is first measured were observed.

ELIGIBILITY:
Inclusion Criteria:

1. patients newly diagnosed with Graves' hyperthyroidism and not treated; or
2. patients diagnosed with Graves' hyperthyroidism and treated with ATDs regularly less than 3 months, serum TSH is measured below normal reference range, serum FT3 or FT4 or both are measured above normal reference range and serum TRAb is positive; or
3. patients diagnosed with Graves' hyperthyroidism and not regularly treated with ATDs more than 3 months, serum TSH is measured below normal reference range, serum FT3 or FT4 or both are measured above normal reference range and serum TRAb is positive.

Exclusion Criteria:

1. thyroid enlargement of grade 3;
2. serum TRAb is measured above 40IU/L;
3. moderate or severe thyroid-associated eye diseases;
4. hepatic disease history including chronic active hepatitis, severe hepatic dysfunction, liver cirrhosis, etc., and serum transaminase level is 3 times higher than the upper normal limit and/or total bilirubin level is higher than 34.2μmol/L with hepatic protective drugs;
5. history of moderate-to-severe or end-stage renal disease: eGFR<60mL/min/1.73m2 with simplified MDRD formula;
6. serum WBC<3.0×109／L or neutrophil count<1.5×109／L;
7. history of severe cardiocerebrovascular disease, digestive disease, hematopoietic system disease, other autoimmune diseases in addition to Graves' hyperthyroidism, tumors, psychosis, etc.;
8. blood pressure>180/100mmHg with regular antihypertensive drugs treatment;
9. severe comorbidities and complications of hyperthyroidism with ATDs treatment;
10. history of multiple drug allergies;
11. a family planning plan in 3 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate of hyperthyroidism | 30 months

SECONDARY OUTCOMES:
Duration from initiation to withdrawal of ATDs | 18 months
Duration from initiation of ATDs to thyroid function (including serum FT3, FT4 and TSH) normalization | 18 months
Duration from initiation of ATDs to serum FT3 and FT4 normalization | 18 months
Quality of life (QOL) in patients with Graves' hyperthyroidism | 30 months
Adverse effects rate of ATDs treatment | 18 months
Duration from initiation of ATDs to serum negative TRAb is first measured | 18 months